CLINICAL TRIAL: NCT03044301
Title: Performance Thresholds Evaluation by Wet Injection Quantification and Magnetic Resonance Imaging (MRI) of Subcutaneous and Intramuscular Injections (0,65ml) of Several Configurations of Needle-free Devices (ZENEO®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crossject (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: G-E-CJT-XC-150127
Record Dates: First submitted 2017-01-09; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: No Condition

ARMS (4):
- BMI < 25kg/m² (Other): Subcutaneous high ZENEO® injection Intramuscular ZENEO® injection
  Interventions: Combination Product: Intramuscular ZENEO® injection; Combination Product: Subcutaneous high ZENEO® injection
- 27.5 > BMI > 25 kg/m² (Other): Intramuscular ZENEO® injection
  Interventions: Combination Product: Intramuscular ZENEO® injection
- BMI > 27.5 kg/m² (Other): Intramuscular ZENEO® injection
  Interventions: Combination Product: Intramuscular ZENEO® injection
- No special BMI (Other): Subcutaneous low ZENEO® injection
  Interventions: Combination Product: Subcutaneous low ZENEO® injection

INTERVENTIONS:
Combination Product: Intramuscular ZENEO® injection — Sodium Chloride (0.9 %)
  Arms: 27.5 > BMI > 25 kg/m²; BMI < 25kg/m²; BMI > 27.5 kg/m²
Combination Product: Subcutaneous high ZENEO® injection — Sodium Chloride (0.9 %)
  Arms: BMI < 25kg/m²
Combination Product: Subcutaneous low ZENEO® injection — Sodium Chloride (0.9 %)
  Arms: No special BMI

SUMMARY:
The aim of this study is to evaluate the performance of the ZENEO needle free device in subcutaneous functioning limits (low performance limit and high performance limit) and for intramuscular injections.

ELIGIBILITY:
Inclusion Criteria:

* male or female healthy volunteers aged between 18 and 60 years,
* affiliated to or covered by the French social security system,
* BMI between ≥20 and ≤30 kg/m²
* Patients without chronic medical or surgical illness
* Patients with normal clinical examination at the screening visit,
* Patients with normal blood pressure at the screening visit: systolic BP < 140 mmHg and diastolic BP < 90 mmHg, determined with the patient seated and resting for at least 5 minutes,
* Patients within normal range values for the following laboratory tests (appendix I) unless the investigator considers an abnormality to be clinically irrelevant (to be documented and agreed with the sponsor before inclusion) within 1 month prior to the start of the study (only for MRI sub study volunteers),
* Absence of cannabis, opiate, cocaine, amphetamine history (only for MRI sub study volunteers)

Exclusion Criteria:

* history of drug abuse
* history of hypersensitivity (disease or drug)
* treatment with platelet inhibiting drugs within one week before inclusion
* treatment with anticoagulant within four weeks before inclusion
* subject likely to take any medication during the study
* contra-indication to MRI: metallic intra-corporeal devices, claustrophobia
* prior participation to other interventional clinical research within 3 months
* in custody due to administrative or legal decision or under tutelage or being admitted in a sanitary or social institution.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
depth of the injection by MRI | 5 minutes after the injection